CLINICAL TRIAL: NCT02749188
Title: Evaluation of Bladder Stimulation as a Noninvasive Technique of Urine Collection in Infants Who Have Not Acquired Walking
Brief Title: Evaluation of Bladder Stimulation as a Noninvasive Technique of Urine Collection in Infant Who Have Not Acquired Walking
Acronym: StiVeN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-HPNCL-07
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-04

CONDITIONS: Urinary Retention
Keywords: Urine Specimen Collection/methods; Infant; Newborn; Feasibility Studies; Bladder stimulation
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bladder stimulation (Other): Bladder stimulation as a noninvasive technique of urine collection. The renal and bladder stimulation will be performed in less than 3 minutes, with a maximum of two attempts spaced about 20 minutes.
  Interventions: Other: Bladder stimulation

INTERVENTIONS:
Other: Bladder stimulation — Bladder stimulation as a noninvasive technique of urine collection. The renal and bladder stimulation will be performed in less than 3 minutes, with a maximum of two attempts spaced about 20 minutes

SUMMARY:
The urinary tract infections are common in children. It is estimated that about 3% of girls and 1% of boys suffer from a urinary tract infection before the age of 11 years. A prompt diagnosis and treatment are necessary for the prevention of morbidity and long-term sequelae.

Currently, there are different methods of urine collection, such as suprapubic aspiration, the survey, the collection bag and the jet medium collection.

They have in common to be time-consuming, invasive in some cases, providers of contaminated levies for others and impossible in children incontinent for the last.

A Spanish study developed a new collection technique, for kidney and bladder stimulation, noninvasive, in the new-born to 30-day months. The results are promising with a success rate of over 85% within a period of about 45s.

No study has looked at a broader pediatric population, including children from birth to age of acquisition of walking.

We hypothesize that it is possible to obtain urine in less than 3 minutes, noninvasively, in infants who have not acquired the works for which a urine sample is required.

DETAILED DESCRIPTION:
The urinary tract infections are common in children. It is estimated that about 3% of girls and 1% of boys suffer from a urinary tract infection before the age of 11 years. A prompt diagnosis and treatment are necessary for the prevention of morbidity and long-term sequelae.

Currently, there are different methods of urine collection, such as suprapubic aspiration, the survey, the collection bag and the jet medium collection.

They have in common to be time-consuming, invasive in some cases, providers of contaminated levies for others and impossible in children incontinent for the last.

A Spanish study developed a new collection technique, for kidney and bladder stimulation, noninvasive, in the new-born to 30-day months. The results are promising with a success rate of over 85% within a period of about 45s.

No study has looked at a broader pediatric population, including children from birth to age of acquisition of walking.

We hypothesize that it is possible to obtain urine in less than 3 minutes, noninvasively, in infants who have not acquired the works for which a urine sample is required.

The main objective is the Evaluation of bladder stimulation as a noninvasive technique of urine collection in infants who have not acquired walking

ELIGIBILITY:
Inclusion Criteria:

* Infants under the age of 2 years and who have not acquired walking
* To which the investigating doctor asked the indication of a urine sample in search of a urinary tract infection, ionic and metabolic disorder
* Do not exhibiting signs of vital distress (respiratory or circulatory or neurological)
* To which the bladder stimulation does not delay the treatment
* Obtaining the authorization of the holders of parental authority
* Affiliation to social security
* Clinical examination

Exclusion Criteria:

* Parental Refusal
* Infants> 2 years or who has walking
* Infant occurring outside the pediatric emergency timetables of care permanently
* Infant having vital signs of distress (respiratory and / or circulatory and / or neurological)
* Infant for which the bladder stimulation could delay the management

Max Age: 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of bladder stimulation as a noninvasive technique of urine collection in infants who have not acquired walking | During baseline at time 0
  • Obtaining urine or not (YES / NO) by bladder stimulation in less than 3 minutes (max 2 attempts). This is evaluated by an investigator who directs the bladder stimulation technique.

SECONDARY OUTCOMES:
evaluation period of urine collection | During baseline at time 0
  If successful, the evaluation period, in seconds, of urine collection using a chronometer (between the start of bladder stimulation and obtaining the urine)
Evaluation of the tolerance of the infant | During baseline at time 0
  Evaluation of the tolerance of the infant undergoing stimulation technique using wide EVENDOL scale pain, noted on 15
alternative of the urine sample | During baseline after 2 attemps of bladder stimulation
  In case of failure, the investigator who included infants in the study will specify the alternative of the urine sample from: collection bag, survey, suprapubic aspiration, and the success or failure of this alternative

CONTACTS AND LOCATIONS:
Overall Officials: Antoine TRAN, MD, Principal Investigator — Fondation Lenval
Locations (1):
- Fondation Lenval, Nice, France

IPD SHARING:
Plan to Share IPD: No